CLINICAL TRIAL: NCT06438692
Title: Clinical Study on the 2C3L Strategy Based on Marshall Venous Chemoablation for the Treatment of Persistent Atrial Fibrillation Combined With Heart Failure
Brief Title: Ablation Strategies for Persistent Atrial Fibrillation Combined With Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05949801
Record Dates: First submitted 2024-01-02; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2C3L group (Sham Comparator): Ablation Procedure：2C3L
  Interventions: Procedure: 2C3L
- 2C3L-plus group (Experimental): Ablation Procedure：2C3L combined with Marshall ethanol ablation
  Interventions: Procedure: VOM ethanol chemical ablation and 2C3L

INTERVENTIONS:
Procedure: VOM ethanol chemical ablation and 2C3L — Annular pulmonary vein ablation, mitral isthmus line ablation, tricuspid isthmus line ablation, apex line ablation，anhydrous alcohol ablation of VOM
  Arms: 2C3L-plus group
Procedure: 2C3L — Annular pulmonary vein ablation, mitral isthmus line ablation, tricuspid isthmus line ablation, apex line ablation
  Arms: 2C3L group

SUMMARY:
(1) To evaluate the efficacy and safety of "2C3L" strategy combined with VOM anhydrous ethanol chemical ablation for persistent atrial fibrillation complicated with heart failure; (2) To evaluate the effectiveness of high-efficiency ablation of atrial fibrillation complicated with heart failure.

DETAILED DESCRIPTION:
2C3L ablation strategy: The electroanatomical mapping system was the Carto 3 V6 system of Johnson & Johnson, and the high-density mapping electrode (Pentaray) and cold saline perfusion pressure catheter (ST-SF) were used for ablation. Ablation parameters were set as follows: ablation power of 45 to 50 Watts (reduced to 25 Watts in the coronary vein and 35 Watts in the endocardium of the mitral isthmus), upper temperature limit of 43 ° C, and saline infusion rate of 15 mL/ min (changed to 30 mL/min in coronary veins), the pressure was controlled at 5-15 g, and the target AI was set: 480-500 for the anterior wall of the pulmonary vein, 350-380 for the posterior wall, 450 for the top of the left atrium, 600 for the mitral valve isthmus, and 450 for the tricuspid valve isthmus. A single catheter procedure was performed in the left atrium, and the ablation endpoint was to achieve continuous bilateral circumferential pulmonary vein damage with loss of intrapulmonary vein potential, which was further confirmed after conversion to sinus rhythm. During left pulmonary vein ablation, the top and posterior wall of left pulmonary vein were ablated first. If pulmonary vein isolation was achieved, no further intervention was performed on the anterior edge of left pulmonary vein. The ablation of the mitral annulus started from about 1 cm away from the junction between the VOM and the coronary vein, and continued to the low-voltage area. Ablation was performed in the corresponding epicardium, namely the coronary vein. Finally, the isthmus of the tricuspid valve was ablated from 6:00 to the inferior vena cava. If the patient still had atrial fibrillation or atrial flutter after the above ablation, 200 J direct current was used to cardioversion the sinus rhythm, and the complete block of each ablation path was verified by pacing during sinus rhythm. In the ablation-only group, catheter ablation was used only to these end points. The operation time was from the start of venipuncture to the removal of sheath tube. The melting time was the cumulative ablation time.

VOM absolute ethanol chemical ablation: The SL1 long sheath was delivered to the opening of the coronary sinus through the right femoral vein, and the right coronary finger guide tube (JR4) was placed to the opening of the coronary sinus. The guide tube was rotated clockwise, and the tip of the guide catheter was pointed in the posterior-superior direction under the right anterior oblique 30 degree fluoroscopy. The BMW guide wire was sent to the proximal end of VOM, and the OTW balloon was sent to the middle and distal end of VOM. The balloon was expanded, and after the BMW guide wire was removed, the course of VOM and whether there was regurgitation were observed by angiography to ensure the complete occlusion of VOM. Anhydrous ethanol was injected in fractions via the OTW balloon.

ELIGIBILITY:
Inclusion Criteria:

1. age:18y-80y
2. First ablation on non valvular atrial fibrillation
3. Persistent atrial fibrillation with LVEF≤40%
4. The patient has symptoms related to atrial fibrillation, including but not limited to palpitations, premonitory syncope, syncope, fatigue, and shortness of breath, and is evaluated for clinical cardiac function between NYHA II-IV levels
5. No response to antiarrhythmic drugs, unacceptable side effects, or unwillingness to take antiarrhythmic drugs.

Exclusion Criteria:

1. Paroxysmal atrial fibrillation
2. Atrial fibrillation secondary to obvious reversible causes
3. Echocardiography: Parasternal long axis section, left atrial diameter ≥ 60mm
4. LVEF >40%
5. Receiving dual antithrombotic therapy
6. Contraindications to the use of oral anticoagulants
7. Contraindications to right or left cardiac catheterization
8. pregnancy
9. Life expectancy<1 year (such as advanced malignant tumors, advanced kidney disease, etc.)
10. Unable to discontinue antiarrhythmic drugs due to reasons other than atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Postoperative recurrence rate | 12 months after operation
  Postoperative recurrence rate was evaluated by holter monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Hu, Study Director — Shandong First Medical University
Locations (1):
- Hesheng Hu, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No